CLINICAL TRIAL: NCT05415592
Title: A Multi-Center, Post-Market, Single-Arm, Observational Clinical Follow-Up Study of Patients Undergoing Radial Head Replacement Using the DePuy Synthes Radial Head Replacement System for Partial Replacement of the Elbow Joint
Brief Title: A Study of Participants Undergoing Radial Head Replacement Using the DePuy Synthes Radial Head Replacement System for Partial Replacement of the Elbow Joint
Status: Withdrawn | Type: Observational
Why Stopped: This was a business decision made due to competing regulatory commitments. Please note that this was not related to the safety or performance of the device.
Sponsor: DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DST202002; DST202002 (Other: DePuy Synthes Products, Inc.)
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Radial Head Fractures
Keywords: Radial Head Replacement; Radial Head Prosthesis; DePuy Synthes,; Partial Elbow Replacement; Device Survivorship
MeSH Terms: conditions — Radial Head and Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- DePuy Synthes Radial Head Replacement System: Participants will undergo a radial head replacement or partial replacement of the elbow joint with the DePuy Synthes Radial Head Replacement System.
  Interventions: Device: DePuy Synthes Radial Head Replacement System

INTERVENTIONS:
Device: DePuy Synthes Radial Head Replacement System — DePuy Synthes Radial Head Replacement System will be used for radial head replacement or partial replacement of the elbow joint.

SUMMARY:
The purpose of this study is to establish survivorship defined by the cumulative incidence of revision over the first 6 months post-implantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female - skeletally mature adult (aged 22 or older)
* Participant, who in the opinion of the Investigator, is able to understand the purpose of the study and is willing to return for all the required post-operative standard of care follow-up visits and have their data collected
* Participant who is willing to give voluntary, written informed consent to participate in this clinical investigation and authorize the transfer of his/her information to the Sponsor

Any one of below:

* Primary replacement after fracture of the radial head
* Participant needing a partial radial head replacement for degenerative or post-traumatic conditions presenting pain, crepitation, and decreased motion at the radio-humeral and/or proximal radio-ulnar joint with: i) joint destruction and/or subluxation visible on x-ray and/or ii. resistance to conservative treatment
* Symptomatic sequelae after radial head resection
* Revision following failed radial head arthroplasty

Exclusion Criteria:

* Dislocations of radius on ulna that would not allow a radio-humeral articulation
* Rheumatoid arthritis
* Infection, sepsis, and osteomyelitis
* Uncooperative participant or participant with neurologic disorders who is incapable of following directions, osteoporosis, metabolic disorders which may impair bone formation, osteomalacia, distant foci of infections which may spread to the implant site, rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Participants with limited life expectancy due to significant medical co-morbidity
* Presence of major vascular or major nerve injury (radial, ulnar, medial, musculocutaneous)
* Women who are pregnant or lactating
* Unable to comply with study requirements example, with maintaining follow-up
* Individuals currently involved in any personal injury litigation, medical-legal or worker's compensation claims
* Individuals that have participated in a clinical investigation with an investigational product (drug or device) in the last three months
* Demented or unable to provide informed consent
* Individuals, in the opinion of the Investigator, who are drug or alcohol abusers or have psychological disorders that could affect their ability to complete participant reported questionnaires or be compliant with follow-up requirements

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include skeletally mature adult participants aged 22 or older who are scheduled to undergo radial head replacement.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Device survivorship Over the First 6 Months Post-implantation | 6 months post-implantation
  Device survivorship is defined by the cumulative incidence of absence of revision. A revision is considered to be any procedure that involves removal of the implant (that is, removal of the Radial Head Prosthesis [RHP], replacement with another RHP or revision surgery to a total elbow arthroplasty).

SECONDARY OUTCOMES:
Number of Participant with Revision Radial Head Replacement (RHR) Surgery | Up to 4 years post surgery
  Number of participants with revision RHR surgery will be reported. Revision surgery reasons include symptomatic aseptic loosening, elbow stiffness, persistent pain, infection, elbow instability, overlengthening, dissociation of the prosthesis, progressive symptomatic ulnohumeral degeneration, secondary fracture, heterotopic ossification, osteoarthritis, erosions of the capitellum, or other implant-related complications.
Assessment of Radiographic Parameters: Mason Classification of Radial Head Fractures | Preoperative, Operative, Discharge (up to Day 6)
  Mason classification system will be used for the classification of radial head fractures. It includes four radial head fracture types. Mason Type I are non-displaced radial head fractures (or small marginal fractures), Mason Type II are partial articular fractures with displacement, Mason Type III are comminuted fractures involving the entire radial head, and Mason Type IV are fractures of the radial head with dislocation of the elbow joint.
Assessment of Radiographic Parameters: Radiolucency | At Months 6, 12, and 24
  Radiolucency will be assessed based on the number of zones involved and the amount of lucency (in millimeters) observed. Radiolucency is classified as: a) None; b) Mild: one or two zones involved by lucent lines of less than (<) 2 millimeters (mm) in thickness; c) Moderate: three to six zones involved or the lucency of greater than or equal to (>=) 2 mm in thickness and d) Severe: all seven zones involved.
Assessment of Radiographic Parameters: Radiocapitellar Alignment | Operative at Week 2, and 6, Months 3, 6, 12, 24, and 48 post operative
  Radiocapitellar alignment will be determined. The position of the radial head prosthesis is assessed on a lateral X-ray based on the intersection between the axis of the prosthetic shaft and the center of the capitellum. The calculation is based on the quotient of the diameter of the trochlea humeri and the axis of the prosthesis.
Assessment of Radiographic Parameters: Ulnohumeral Degeneration | Operative at Week 2, and 6, Months 3, 6, 12, 24, and 48 post operative
  Ulnohumeral degeneration will be assessed. The degree of ulnohumeral degeneration is classified with the system described by Broberg and Morrey as Grade 0 (normal joint), Grade 1 (slight joint space narrowing with minimum osteophyte formation), Grade 2 (moderate joint space narrowing with moderate osteophyte formation) or Grade 3 (severe degenerative changes with gross destruction of the joint).
Assessment of Radiographic Parameters: Osteoarthritis | At Week 2, and 6, Months 3, 6, 12, 24, and 48
  Osteoarthritis (in the radio-capitellar joint) will be assessed. Osteoarthritis is evaluated as yes/no, if yes, the location will be described (that is., medial, lateral or both).
Assessment of Radiographic Parameters: Heterotopic Ossification | At Week 2, and 6, Months 3, 6, 12, 24, and 48
  Heterotopic ossification will be determined and reported. Heterotopic ossification is classified as present (that is, anterior-posterior, medial-lateral) or absent.
Assessment of Radiographic Parameters: Osteopenia, and/or Capitellar Abrasion | At Week 2, and 6, Months 3, 6, 12, 24, and 48
  Osteopenia, and/or capitellar abrasion will be determined and reported. Capitellar osteopenia and/or abrasion is classified as none, mild, moderate, or severe.
Assessment of Radiographic Parameters: Overlengthening | Operative at Months 6, 12, and 24 post operative
  Overlengthening will be determined and reported. Overlengthening is assessed on the intra- or postoperative, 6-, 12- and 24 months Antero-Posterior (AP) and lateral X-rays (evidence of overstuffing).
Assessment of Radiographic Parameters: Joint incongruity | Operative at Week 2, and 6, Months 3, 6, 12, 24 and 48 post operative
  Joint incongruity will be determined and reported. Joint incongruity is assessed as yes/no.
Mayo Elbow Performance Index (MEPI) Score | Week 2 and 6, Months 3, 6, 12, 24, and 48
  MEPI is also known as Mayo Elbow Performance Score (MEPS). MEPI is used to evaluate the clinical outcomes for a variety of elbow disorders such as elbow fractures and dislocations. The MEPI is a validated hundred-point system based upon pain (forty five points), range of motion (twenty points), stability (ten points) and daily function (twenty five points) The scale ranges from 0 to 100, with a higher score indicating a better outcome.
Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) Score | Week 2 and 6, Months 3, 6, 12, 24, and 48
  QuickDASH questionnaire has 30-items, which includes 21 items for physical function, 6 for symptoms, and 3 for social roles. Quick DASH is a shorter version, developed for less burden to the responder. It consists of 11 items out of the original 30 questions of the DASH. QuickDASH is scored between 0 (no disability) to 100 (most severe disability), with lower scores indicating better overall wellness.
Elbow Range of Motion (ROM) | Week 2 and 6, Months 3, 6, 12, 24, and 48
  Elbow ROM of both sites (injured side and contralateral side) will be assessed according to standard of care practices for elbow flexion, elbow extension, forearm supination, and forearm pronation.
Grip Strength of the Injured Limb Compared to the Contralateral Side | At Week 6, Months 6, 12, 24 and 48
  The grip strength (if available) will be assessed with dynamometer following the standardized testing protocol recommended by the American Society of Hand Therapists (ASHT). For measurements, the participants would be in a comfortable sitting position in a chair without arm rests, with feet fully resting on the floor, hips as far back in the chair as possible, and the hips and knees positioned at approximately 90 degrees. Grip force should be applied smoothly, without rapid wrenching or jerking motion. (No correction for hand dominance will be performed because this effect varies substantially among users. Assessment will be also performed on the unaffected side using the same method.
European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Scale Score | Preoperative, Week 6, Months 6, 12, 24, and 48
  EQ-5D-5L questionnaire includes five questions (descriptive system: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a visual analog scale to rate the current health status. The resulting scores were converted into a single index score that ranged from -0.281 to 1, where higher score indicates better health. Values lower than 0 represent states considered to be worse than death.
Local Pain Assessed by Numerical Rating Scale (NRS) Score | Week 2 and 6, Months 3, 6, 12, 24, and 48
  Local pain intensity levels over the previous 24 hours will be assessed with the Numerical Rating Scale (NRS). The scale range goes from 0 (no pain) to 10 (worst imaginable pain). A higher value correlates with greater pain.
Number of Participants who Return to Work and Sport | Week 2 and 6, Months 3, 6, 12, 24, 36 and 48
  Number of participants who return to work and Sport will be assessed as yes/no.
Number of Participants with Device and/or Procedure-related Adverse Events (AEs) | Operative, Discharge (up to Day 6), Week 2, 6, Months 3, 6, 12, 24, 36, and 48
  Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, users or other persons, whether or not related to investigational medical device, the Radial Head Replacement System, and whether anticipated or unanticipated.
Number of Participants with Device and/or Procedure-related Serious Adverse Events (SAEs) | Operative, Discharge (up to Day 6), Week 2, 6, Months 3, 6, 12, 24, 36, and 48
  SAEs are defined as any device and or procedure related adverse event that: 1. Led to death; 2. Serious deterioration in the health of the subject, that resulted in any of the following: a. life-threatening illness or injury, b. permanent impairment of a body structure or a body function, c. hospitalization or prolongation of existing hospitalization, d. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function, e. chronic disease; 3. Led to fetal distress, fetal death or a congenital physical or mental impairment or birth defect.
Number of Participants with Revision/Reoperations | Operative, Discharge (up to Day 6), Week 2, 6, Months 3, 6, 12, 24, 36, and 48
  Number of participants with revision/reoperation will be reported. A revision is considered to be any procedure that involves removal of the implant (that is, removal of the RHP, replacement with another RHP or revision surgery to a total elbow arthroplasty). Reoperation is defined as a second operation involving the DePuy Synthes Radial Head Replacement System at the index site and after the index surgery that does not include removal or replacement of the implanted Radial Head Prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: DePuy Synthes Products, Inc. Clinical Trial, Study Director — DePuy Synthes Products, Inc.
Locations (4):
- United States (3):
  - MetroHealth Medical Center, Cleveland, Ohio
  - Slocum Research & Education Foundation, Eugene, Oregon
  - Inova Orthopaedics - Fairfax, Falls Church, Virginia
- Glasgow Royal Infirmary (NHS Greater Glasgow & Clyde), Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agyeman KD, Damodar D, Watkins I, Dodds SD. Does radial head implant fixation affect functional outcomes? A systematic review and meta-analysis. J Shoulder Elbow Surg. 2019 Jan;28(1):126-130. doi: 10.1016/j.jse.2018.07.032. Epub 2018 Oct 17. PMID 30342823
- [Background] Bahreini M, Safaie A, Mirfazaelian H, Jalili M. How much change in pain score does really matter to patients? Am J Emerg Med. 2020 Aug;38(8):1641-1646. doi: 10.1016/j.ajem.2019.158489. Epub 2019 Nov 4. PMID 31744654
- [Background] Bain, G., Eygendaal, D., and van Riet, R. (2020). Surgical Techniques for Trauma and Sports Related Injuries of the Elbow
- [Background] Broberg MA, Morrey BF. Results of delayed excision of the radial head after fracture. J Bone Joint Surg Am. 1986 Jun;68(5):669-74. PMID 3722222
- [Background] Churchill RW, Munoz J, Ahmad CS. Osteochondritis dissecans of the elbow. Curr Rev Musculoskelet Med. 2016 Jun;9(2):232-9. doi: 10.1007/s12178-016-9342-y. PMID 27125506
- [Background] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787
- [Background] Cusick MC, Bonnaig NS, Azar FM, Mauck BM, Smith RA, Throckmorton TW. Accuracy and reliability of the Mayo Elbow Performance Score. J Hand Surg Am. 2014 Jun;39(6):1146-50. doi: 10.1016/j.jhsa.2014.01.041. Epub 2014 Mar 20. PMID 24656392
- [Background] Devlin NJ, Shah KK, Feng Y, Mulhern B, van Hout B. Valuing health-related quality of life: An EQ-5D-5L value set for England. Health Econ. 2018 Jan;27(1):7-22. doi: 10.1002/hec.3564. Epub 2017 Aug 22. PMID 28833869
- [Background] Duckworth AD, McQueen MM, Ring D. Fractures of the radial head. Bone Joint J. 2013 Feb;95-B(2):151-9. doi: 10.1302/0301-620X.95B2.29877. PMID 23365021
- [Background] Fowler JR, Goitz RJ. Radial head fractures: indications and outcomes for radial head arthroplasty. Orthop Clin North Am. 2013 Jul;44(3):425-31, x. doi: 10.1016/j.ocl.2013.03.013. Epub 2013 Apr 17. PMID 23827844
- [Background] Gao Y, Zhang W, Duan X, Yang J, Al-Qwbani M, Lv J, Xiang Z. Surgical interventions for treating radial head fractures in adults. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD008987. doi: 10.1002/14651858.CD008987.pub2. PMID 23728684
- [Background] Gerbershagen HJ, Rothaug J, Kalkman CJ, Meissner W. Determination of moderate-to-severe postoperative pain on the numeric rating scale: a cut-off point analysis applying four different methods. Br J Anaesth. 2011 Oct;107(4):619-26. doi: 10.1093/bja/aer195. Epub 2011 Jun 30. PMID 21724620
- [Background] Giannicola G, Sacchetti FM, Antonietti G, Piccioli A, Postacchini R, Cinotti G. Radial head, radiocapitellar and total elbow arthroplasties: a review of recent literature. Injury. 2014 Feb;45(2):428-36. doi: 10.1016/j.injury.2013.09.019. Epub 2013 Sep 19. PMID 24112701
- [Background] GmbH, S. (2020). Instructions for Use - Radial Head Replacement System (https://ifu.depuysynthes.com/?lang=en&archive=&keyword=Radial+Head).
- [Background] Grewal R, MacDermid JC, Faber KJ, Drosdowech DS, King GJ. Comminuted radial head fractures treated with a modular metallic radial head arthroplasty. Study of outcomes. J Bone Joint Surg Am. 2006 Oct;88(10):2192-200. doi: 10.2106/JBJS.E.00962. PMID 17015596
- [Background] Gummesson C, Atroshi I, Ekdahl C. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: longitudinal construct validity and measuring self-rated health change after surgery. BMC Musculoskelet Disord. 2003 Jun 16;4:11. doi: 10.1186/1471-2474-4-11. Epub 2003 Jun 16. PMID 12809562
- [Background] Heijink A, Kodde IF, Mulder PGH, Veltman ES, Kaas L, van den Bekerom MPJ, Eygendaal D. Radial Head Arthroplasty: A Systematic Review. JBJS Rev. 2016 Oct 18;4(10):e3. doi: 10.2106/JBJS.RVW.15.00095. PMID 27792673
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Jung M, Groetzner-Schmidt C, Porschke F, Grutzner PA, Guehring T, Schnetzke M. Low return-to-sports rate after elbow injury and treatment with radial head arthroplasty. J Shoulder Elbow Surg. 2019 Aug;28(8):1441-1448. doi: 10.1016/j.jse.2019.03.014. Epub 2019 Jun 18. PMID 31227468
- [Background] Kaas L, van Riet RP, Vroemen JP, Eygendaal D. The epidemiology of radial head fractures. J Shoulder Elbow Surg. 2010 Jun;19(4):520-3. doi: 10.1016/j.jse.2009.10.015. Epub 2010 Feb 10. PMID 20149972
- [Background] Lamas C, Castellanos J, Proubasta I, Dominguez E. Comminuted radial head fractures treated with pyrocarbon prosthetic replacement. Hand (N Y). 2011 Mar;6(1):27-33. doi: 10.1007/s11552-010-9282-8. Epub 2010 Jun 15. PMID 22379435
- [Background] Lapner M, King GJ. Radial head fractures. J Bone Joint Surg Am. 2013 Jun 19;95(12):1136-43. No abstract available. PMID 23943926
- [Background] MacDermid, J., Solomon, G., Valdes, K., and American Society of Hand, T. (2015). Clinical assessment recommendations
- [Background] Mansat P. Surgical treatment of the rheumatoid elbow. Joint Bone Spine. 2001 May;68(3):198-210. doi: 10.1016/s1297-319x(01)00273-1. PMID 11394619
- [Background] Merolla G, Buononato C, Chillemi C, Paladini P, Porcellini G. Arthroscopic joint debridement and capsular release in primary and post-traumatic elbow osteoarthritis: a retrospective blinded cohort study with minimum 24-month follow-up. Musculoskelet Surg. 2015 Sep;99 Suppl 1:S83-90. doi: 10.1007/s12306-015-0365-0. Epub 2015 May 10. PMID 25957550
- [Background] Murphy, A. Elbow (Coyle's view) (Radiopaedia)
- [Background] Skytta ET, Eskelinen A, Paavolainen P, Ikavalko M, Remes V. Total elbow arthroplasty in rheumatoid arthritis: a population-based study from the Finnish Arthroplasty Register. Acta Orthop. 2009 Aug;80(4):472-7. doi: 10.3109/17453670903110642. PMID 19562563
- [Background] Synthes, D. (2020a). Instructions for Use - Radial Head Replacement System
- [Background] Synthes, D. (2020b). Radial Head Replacement System Surgical Technique
- [Background] Synthes, D. (2020c). Radial Head Replacement System Surgical Technique Guide, pp. Surgical Technique Guide
- [Background] Tarallo L, Mugnai R, Rocchi M, Capra F, Catani F. Mason type III radial head fractures treated by anatomic radial head arthroplasty: Is this a safe treatment option? Orthop Traumatol Surg Res. 2017 Apr;103(2):183-189. doi: 10.1016/j.otsr.2016.10.017. Epub 2016 Dec 8. PMID 27940249